CLINICAL TRIAL: NCT05516849
Title: Placebo Versus Oxandrolone Supplementation in Trauma: A Randomized Multi-Center Double Blind Clinical Trial in High-Energy Lower Extremity Trauma (POST-Injury Trial)
Brief Title: Placebo Versus Oxandrolone Supplementation in Trauma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: FDA requested manufacturers of Oxandrolone Tablets, to voluntarily remove previously approved drug applications for Oxandrolone from the U.S. market & the funding decided to prematurely terminate the funding.
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3822: POST-INJURY
Record Dates: First submitted 2022-08-16; First posted 2022-08-26 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Trauma Injury
MeSH Terms: conditions — Accidental Injuries | interventions — Oxandrolone

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 fashion to one of the two treatment arms using a minimal sufficient randomization technique in REDCAP.
Who Masked: Participant, Investigator
Masking Description: All participants, clinicians, and staff will be blinded to the intervention groups. All patients with an adverse event will be reviewed by an onsite internal medicine affiliated with the study but not directly in recruitment or assessment of outcomes. Emergency unblinding will be allowed if participants present with an adverse event that in the opinion of consulting physicians is not explained by other causes AND knowing the treatment allocation will aid in the patient's management. The blind may be broken only with the permission of the Principal Investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oxandrolone (Experimental): Participants will be randomly assigned in a 1:1 fashion to one of the two treatment arms using the REDCap database randomization procedure.
  Interventions: Drug: Oxandrolone
- Placebo (Placebo Comparator): Participants will be randomly assigned in a 1:1 fashion to one of the two treatment arms using the REDCap database randomization procedure.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oxandrolone — Oxandrolone is a synthetic anabolic androgenic steroid that induces its responses by binding to androgen receptors which modulates gene expression to increase protein synthesis and efficient utilisation of amino acids. Oxandrolone was first synthesized in 1962 through 17alpha-alkylation of testosterone resulting in a formal composition of (4bS,7S,9aS,9bR,11aS)-tetradecahydro-7-hydroxy-4aS,6aS,7-trimethyl- cyclopentanaphthopyran-2(1H)-one and molecular formula of C19H30O3.
  Arms: Oxandrolone
Other: Placebo — As there is currently no approved medication to aid in soft-tissue regeneration, we will be using a placebo control.
  Arms: Placebo

SUMMARY:
The primary aim of this study is to examine the effect of Oxandrolone supplementation after lower extremity high energy fracture on muscle volume recovery. As Oxandrolone supplementation has never been examined in this patient population, the primary null hypothesis is that there will be no difference in measured thigh muscle mass volume between Oxandrolone supplementation and placebo administration groups.

DETAILED DESCRIPTION:
Lower extremity fractures associated with high-energy mechanisms of injury (combat injuries including blast or crush injuries, motor vehicle accidents, fall from significant height, gunshot injuries) are unfortunately common among active service members and civilians presenting to level-1 trauma centers worldwide. High-energy fractures have several unique characteristics that distinguish them from low-energy injuries. They typically occur in predominately younger, male patients (30-65 years old)1 and involve significant soft-tissue stripping or damage. These patients require at least one major reconstructive surgery, with the majority requiring multiple reconstructive surgeries, each associated with additional soft tissue injury and subsequent prolonged immobilization to facilitate limb stabilization. Despite extended rehabilitation focused on neuromuscular retraining and muscular development, the result is often permanent limitations of ambulation and medical retirement from active duty due to volumetric muscle loss. So, while advances in orthopedic approaches to fracture care have lowered complications such as non-union and malunion, rendering them less significant as limitations to restoring function soft-tissue complications now predominate.

Oxandrolone has been successfully utilized to accelerate muscular recovery, reduce muscle loss, and improve function in several populations including healthy elderly patients with frailty/sarcopenia, patients with large surface area burns, neuromuscular diseases, HIV, congenital heart disease and genetic diseases including Klinefelter's and Turner's Syndromes. In addition, Oxandrolone has also been safely used in pediatric patients to treat constitutionally delayed growth. Given the similarities in patient populations and the known limitations of volumetric muscle loss in military personnel and civilians after major trauma, Oxandrolone supplementation may reduce initial volumetric muscle loss and improve long-term muscle mass and function.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Ages 18-55 [inclusive]
3. Skeletally-mature as based upon tibial or femoral physeal closure41
4. Fracture of the femur or tibia treated with open reduction and internal fixation (simple articular patterns allowed).
5. High energy injuries with associated local soft tissue damage. -

Exclusion Criteria:

1. Unable to participate in rehabilitation including severe head injury, pre-existing TBI or cognitive dysfunction (stroke, dementia, documented developmental delay), patients with significant spinal cord injury or pre-accident paralytic injury or condition will beessential treatment in both intervention and control groups.
2. Medically unfit for anabolic steroid treatment including those with active malignancy, concurrent prednisone use, elevated liver enzymes at baseline (baseline bloodwork to include LFT)
3. Fracture due to primary or metastatic bone lesion
4. Any contraindications to MRI.
5. Patients with major psychiatric illness [trauma presentation for suicide attempts] and incarcerated patients will be excluded as they may lack autonomy, decision-making capacity and the ability to meet follow-ups.
6. Patients with substance use disorders, due to increased abuse potential and possible baseline hepatic injury.
7. Patients who are on blood thinning medication, at baseline.
8. Patients receiving hormone treatment.
9. Patients with active cancers.
10. Patients with a history of hypercalcemia/parathyroid disease and chronic renal disease.

    -

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2022-05-19 (Estimated); Primary Completion 2023-08-03 (Estimated); Study Completion 2023-08-03 (Estimated)

PRIMARY OUTCOMES:
Delta volumetric vastus medialis diameter on MRI | upto 6 months
  MRI is taken to assess the vastus medialis muscle mass.

SECONDARY OUTCOMES:
Delta volumetric thigh muscle mass on MRI | Up to 1 year
  Delta volumetric thigh muscle mass on MRI at 52 week Post treatment and the VMO (Vastus Medialis) at 26 week visit.
Functional measure: 6-minute walk test | Up to 1 year
Activity count by ActiGraph GT3X-BT | Up to 1 year
  The actigraph measures sleep efficiency.
Short Form 36 Health Survey | Up to 1 year
  The minimum score is 0, and maximum score is 5.
Patient-Reported Outcomes Measurement Information System (PROMIS) | Up to 1 year
  The minimum score is 0, and maximum score is 10.
Standard AP and Lateral X-Rays | Through study completion, an average of 1 year
  Time to radiographic union of fracture in weeks based on bridging callous of 3 of 4 cortices on standard AP and lateral x-rays
Length of in-patient Acute Hospital stay, and Rehabilitation stay | Through study completion, an average of 1 year
  Length of in-patient Acute Hospital stay, and Rehabilitation stay to be determined by the orthopedic surgeon.
MARX Scale | Up to 1 year
  The minimum score is 0, and maximum score is 10.
VAS Score | Up to 1 year
  The minimum score is 0, and maximum score is 10.
Hand-Held Dynamometer | Up to 1 year
  The hand-held dynamometer is a small device that fits in the examiner's hand and is placed at precise locations on a subject's limb in an effort to assess the force generated by various muscles or groups of muscles.The minimum score is 0, and maximum score is 10.

IPD SHARING:
Plan to Share IPD: No